CLINICAL TRIAL: NCT04238871
Title: Idiopathic Interstitial Pneumopathy : Genetic and Environmental Determinants From Infancy to Elderly
Brief Title: RaDiCo PID Cohort (RaDiCo-ILD Cohort in English)
Acronym: RaDiCo-PID
Status: Recruiting | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C15-64
Record Dates: First submitted 2019-11-25; First posted 2020-01-23 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Idiopathic Interstitial Pneumopathy/Pneumopathy Interstitial Diffuse; Paediatric and Adult Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- children or adults with Idiopathic Lung Disease

SUMMARY:
The main objective is to describe the phenotypic features of the paediatric and adult patients with Idiopathic Interstitial Pneumopathy/Pneumopathy Interstitial Diffuse (IIP/PID), at diagnosis and during the follow-up. These data will be critical for the description of the natural history of the various forms of IIP/PID.

DETAILED DESCRIPTION:
The French RaDiCo-PID : Idiopathic Interstitial Pneumopathy registry is an ongoing observational prospective and retrospective cohort with longitudinal long-term follow-up includes pediatric and adult patients with Idiopathic Interstitial Lung Disease (ILD) from the reference and competence centers.

ELIGIBILITY:
Inclusion Criteria:

* Clinical criteria: chronic respiratory insufficiency manifestations including dyspnea/tachypnea, cough, and cyanosis during exercise or at rest
* Radiological criteria: characteristic chest High-Resolution Computed Tomography (HRCT) abnormalities including widespread ground glass or alveolar attenuation, reticulation often associated with traction bronchiectasis, and honeycombing
* Functional criteria: pulmonary function test abnormalities reflecting a restrictive pattern and including: loss of lung volume, vital capacity (VC), total lung capacity (TLC); reduction in the diffusion capacity of the lung for carbon monoxide (DLCO), gas exchange abnormalities, and altered ventilatory response to exercise
* Patients (parents/guardians for paediatric/patients) having given an informed consent to participate in the protocol
* Patients affiliated to the "Regime National d'Assurance Maladie"

Exclusion Criteria:

* Patients with diffuse parenchymal lung diseases caused by drug toxicity, immunodeficiency, proliferative disorders including histiocytosis, and metabolic disorders
* Patients (parents/guardians for paediatric patient) not able to approve/understand the protocol

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient with a diagnosis of Pneumopathie Interstitielle Diffuse/ Idiopathic Interstitial Pneumonia diagnosis is established on presenting history, clinical, radiological and functional and if available pathological findings.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2017-06-21 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The phenotypic description idiopathic lung disease | Up to 10 years
  Phenotypic description will be measure demographic data, environmental data, socio-professionnal data, medical history, comorbidities, clinical examination, biological assessment (hematology; biochemistry; hemostasis...), pulmonary biopsy, bronchial-pulmonary imaging; symptom description; respiratory function (arterial blood gas, pulmonary fonction testing, six minute-walk testing, cardiopulmonary exercise testing, polysomnography), treatments, quality of life questionnaire (SF36 and SF10)

SECONDARY OUTCOMES:
Identify gene factors involved in disease initiation and progression | Up to 10 years
  study genes : SFTPA1, SFTPA2, SFTPB, SFTPC, ABCA3, NKX-2.1, TERT, TERC, RTEL1, PARN, DKC1, TINF2, COPA, MARS, CSF2RA, CSF2RB, SERPINA1, FLCN
Investigate the extent to which environmental and co-morbidity factors may influence disease severity and outcome | Up to 10 years
  environnemental data: dwellings, wet areas, dust, smoking, drugs, exposure to materials. Respiratory history, cardiovascular history, endocrinal history, dermatological history, gastroenterology history, gynecology history, haematological history, immune history, neurological history, ophtalmological history, ENT history, psychatric history, Rheumatology history, surgery history
Identify and validate biomarkers for disease diagnosis and progression | Up to 10 years
  Identify and validate biomarkers for disease diagnosis and progression with Biological assessment (professionnal data, medical history, comorbidities, clinical examination, biological assessment (hematology; biochemistry; hemostasis...) and respiratory function (arterial blood gas, pulmonary fonction testing, six minute-walk testing, cardiopulmonary exercise testing, polysomnography)

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU Lyon - Hôpital Louis Pradel, Bron
  - AP-HP - Hôpital Armand Trousseau, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cottin V, Gueguen S, Nunes H, Jouneau S, Crestani B, Bonniaud P, Wemeau L, Israel-Biet D, Reynaud-Gaubert M, Gondouin A, Cadranel J, Marchand-Adam S, Chevereau M, Dufaure-Gare I, Amselem S, Clement A; and the RaDiCo team. Treatment of Idiopathic Pulmonary Fibrosis with Capsule or Tablet Formulations of Pirfenidone in the Real-Life French RaDiCo-ILD Cohort. Adv Ther. 2022 Jan;39(1):405-420. doi: 10.1007/s12325-021-01961-x. Epub 2021 Nov 10. PMID 34757602